CLINICAL TRIAL: NCT05253131
Title: Phase 1/2 Trial of the MEK Inhibitor Selumetinib and Bromodomain Inhibitor ZEN-3694 With Durvalumab (MEDI4736), a PD-L1 Antibody for Sarcomas Including Malignant Peripheral Nerve Sheath Tumors
Brief Title: Trial of Selumetinib and Bromodomain Inhibitor With Durvalumab for Sarcomas
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Girish Dhall, MD, PI, NFCTC, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 300006373; W81XWH-17-2-0037 NF160012 (Other Grant/Funding Number: DoD - Congressionally Directed Medical Research Program)
Record Dates: First submitted 2022-02-03; First posted 2022-02-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: MPNST; NF1; Sarcoma
Keywords: MPNST; Neurofibromatosis 1; NF1; sarcoma
MeSH Terms: conditions — Neurofibrosarcoma; Sarcoma; Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Intervention Model Description: Part A will be a phase 1 dose escalation study of the combination with selumetinib and BI.
  Part B will be phase 1 study combining the determined dose of selumetinib and BI from Part A with durvalumab.
  Part C will be a phase 2 study combining selumetinib, BI with durvalumab in MPNST patients at the recommended doses from part B. A Simon's two-stage design will be used in the phase 2 trial to determine the clinical benefit in patients with unresectable or metastatic NF associated MPNST.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 and 2 Study of Selumentinib, ZEN-3694 and Durvalumab (Experimental): Part A will be a phase 1 dose escalation study of the combination with selumetinib and ZEN-3694.
  Part B will be phase 1 study combining the determined dose of selumetinib and ZEN-3694 from Part A with durvalumab.
  Part C will be a phase 2 study combining selumetinib, ZEN-3694 with durvalumab in MPNST patients at the recommended doses from part B. A Simon's two-stage design will be used in the phase 2 trial to determine the clinical benefit in patients with unresectable or metastatic NF associated MPNST.
  Interventions: Combination Product: Selumetinib + ZEN-3694 ± Durvalumab

INTERVENTIONS:
Combination Product: Selumetinib + ZEN-3694 ± Durvalumab — Selumetinib and ZEN-3694 administered per protocol, with durvalumab added in later study parts.

SUMMARY:
A multi-institutional open-label phase 1/2 trial of selumetinib in combination with ZEN-3694 and durvalumab in refractory/unresectable sarcomas including MPNST. The phase 1 portion will be separated in two parts and will be open to all patients with refractory/relapsed sarcomas. The phase 2 portion will be for patients with refractory/unresectable NF1-associated MPNST.

DETAILED DESCRIPTION:
A multi-institutional open-label phase 1/2 trial of selumetinib in combination with bromodomain inhibitor (ZEN-3694) and durvalumab in refractory/unresectable sarcomas including MPNST. The phase 1 portion will be separated in two parts and will be open to all patients with refractory/relapsed sarcomas. The phase 2 portion will be for patients with refractory/unresectable NF1-associated MPNST.

Part A will be a phase 1 dose escalation study of the combination with selumetinib and ZEN-3694.

Part B will be phase 1 study combining the determined dose of selumetinib and ZEN-3694 from Part A with durvalumab.

Part C will be a phase 2 study combining selumetinib, ZEN-3694 with durvalumab in MPNST patients at the recommended doses from part B. A Simon's two-stage design will be used in the phase 2 trial to determine the clinical benefit in patients with unresectable or metastatic NF associated MPNST.

Statistical Plan Phase 1: Conventional dose escalation schema. Cohorts of 3 to 6 participants will be treated per dose level. At the RP2D or last dose level, the cohort may be expanded to up to an additional six participants for further pharmacokinetic and tolerability experience. The MTD/RP2D will be defined as the dose level immediately below the level at which ≥33% of participants in a cohort experience a DLT based on toxicities observed in the first drug therapy cycle.

Phase 2: A Simon's two-stage phase 2 trial of selumetinib, ZEN-3694, and durvalumab to determine the safety and clinical benefit in patients with unresectable or metastatic MPNST Maximum Total Number of Subjects Phase 1: 6-24 participants Phase 2: 9 participants in first stage with additional 8 participants in stage 2.

Target Population Individuals ≥ 18 years of age with relapsed or refractory histologically confirmed sarcoma including MPNST. This may be amended when tolerability is established.

Anticipated Length of Study Maximum enrollment number for entire study is 41participants. It is expected that 15-25 participants will be enrolled per year, and enrollment is expected to be completed in 3 years with follow up after last participant accrual to be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria AGE: ≥ 18 years of age Weight: >30 kg Life expectancy of at least 12 weeks

Part A and B (Phase 1): Patients with histologically confirmed soft tissue or bone sarcoma of the following subtypes:

* MFH/ undifferentiated pleomorphic sarcoma
* Unclassified sarcoma
* Rhabdomyosarcoma
* Malignant peripheral nerve sheath tumor (MPNST)
* Osteosarcoma
* Ewing or Ewing-like sarcoma
* Synovial sarcoma
* Desmoplastic small round blue cell tumor (DSRCT)

Patients must have progressed or demonstrated disease that is refractory to standard therapies.

Patients for whom no standard of care treatments exist are eligible.

Part C (Phase 2): Patients with progressive, relapsed, unresectable or metastatic NF associated MPNST.

MEASURABLE DISEASE:

Patients must have evaluable or measurable disease (Phase 1) and measurable disease by RECISTv1.1 (Phase 2).

* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study excluding chronic grade 1 toxicities and alopecia.
* No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.
* Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks (≥21 days) and 42 days if prior nitrosourea prior to study entry.
* Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.
* Biologic (anti-cancer agent): The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry. Prior therapy with a MEK, Ras, or Raf inhibitor used for treatment of malignant sarcoma is not allowed. Prior therapy of MEK, Ras, or Raf inhibitor for other tumor such as plexiform neurofibroma or glioma is allowed.
* Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study
* Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.
* Stem Cell Transplantation. At least 2 months post-autologous stem cell transplant.
* Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.
* Karnofsky performance level ≥ 50% (See Appendix II).
* Patients who are unable to walk because of paralysis or motor weakness, but who are able to use a wheelchair will be considered ambulatory for the purpose of calculating the performance score.

Hemoglobin ≥9.0 g/dL (transfusion permissible)

* Peripheral absolute neutrophil count (ANC) of ≥1000/µL
* Platelet count ≥100,000/µL (transfusion independent (no transfusion within at least 7 days prior to enrollment))
* Total bilirubin must be ≤ 1.5 times the upper limit of normal (ULN)
* SGOT (AST)/SGPT (ALT) must be ≤ 3.0 times ULN unless liver metastases are present, in which case it must be ≤ 5x ULN

RENAL FUNCTION:

Serum creatinine ≤ 1.5 times ULN or measured reatinine clearance >50 mL/min or calculated creatinine clearance > 50 mL/min by the Cockcroft- Gault formula (Cockgraft and Gault 1976) or by the 24 hour urine collection for determination of creatinine clearance

* Normal ejection fraction (ECHO or cardiac MRI) ≥53% (or the institutional normal; if a range is given then the upper value of the range will be used)
* QTC or QTcF ≤ 450msec

Fertile men and women of childbearing potential must agree to use an effective method of birth control.

Female participants of childbearing potential must be willing to practice highly effective contraception as detailed below from the time of screening until 3 months after discontinuing the study.

They must not be breastfeeding and must have negative pregnancy test prior to start of dosing.

For a female participant to be considered as of not childbearing potential, she should fulfil one of the following:

Post-menopausal women, defined as either women aged more than 50 years and have amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments, or, women under 50 years who have amenorrhea for at least 12 months following cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels in the postmenopausal range for the institution.

or

* Have documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (but not tubal ligation)
* Have medically confirmed, irreversible premature ovarian failure.

Highly effective methods of contraception are:

* Use of medroxyprogesterone acetate depot injection (Depo-proveraTM). (Please note: use of any other oral, injected, or implanted hormonal methods of contraception cannot be considered highly effective as it is currently unknown whether investigational agents may reduce their effectiveness)
* Placement of a copper-banded intrauterine device (IUD) or intrauterine system (IUS)
* Bilateral tubal ligation
* Vasectomized partner

Barrier methods include:

Occlusive cap (e.g. diaphragm or cervical/vault caps) with spermicide

Male participants should either be surgically sterile or willing to use an effective barrier method of contraception during the study and for 3 months following the last dose of drug therapy if sexually active with a female of childbearing potential. If not done, storage of sperm prior to receiving drug therapy will be advised to male participants with a desire to have children.

Male subjects must agree to refrain from sperm donation during and until 90 days from drug therapy discontinuation.

CNS DISEASE: Patients with central nervous system disease are eligible or enrollment if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of clinical progression or stable disease at 4 weeks.

Exclusion Criteria:History of another primary malignancy except for

* A malignancy treated with curative intent and with no known active disease ≥5 years prior to study entry
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* Stable optic pathway glioma or low grade glioma not receiving active therapy

History of leptomeningeal carcinomatosis.

Patients receiving other anti-cancer agents are not eligible.

Patients who cannot swallow whole pills.

History of allogeneic organ transplantation.

Current or prior use of immunosuppressive medications within 14 days prior to study entry. The following are exceptions to this criterion:

intranasal, inhaled, topical steroids or local steroid injection (e.g., intra-articular injection)

Systemic corticosteroids used at physiologic doses not to exceed 10mg/day of prednisone or its equivalent.

Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).

Patients should not receive immunizations with attenuated live vaccines within four weeks of study entry or during study period.

Any recent major surgery within a minimum of 4 weeks prior to starting drug therapy. Placement of vascular access device, percutaneous tumor biopsy, or bone marrows are not considered major surgical procedures and no minimum time frame prior to starting study drug.

Patients who have any known severe and/or uncontrolled medical therapy is required.

conditions or other conditions that could affect their participation in the study such as:

* Severely impaired lung function defined as spirometry and DLCO that is 50%of the normal predicted value corrected for hemoglobin and alveolar volume and/or O2 saturation that is 88% or less at rest on room air. For patients who do NOT have respiratory symptoms (e.g., dyspnea at rest, known requirement for supplemental oxygen), pulmonary function test is not required.
* Cardiac conditions as follows:

  * Uncontrolled hypertension (blood pressure ≥150/95 mmHg despite medical therapy.
  * Acute coronary syndrome within 6 months prior to starting drug therapy
  * Uncontrolled angina despite medical therapy (Canadian Cardiovascular Society grade II-IV despite medical therapy
  * Symptomatic heart failure NYHA Class II-IV prior or current cardiomyopathy or severe valvular disease
  * Prior or current cardiomyopathy including but not limited to the following: Known hypertrophic cardiomyopathy; Known arrhythmogenic right ventricular cardiomyopathy; or Previous moderate or severe impairment of left ventricular systolic function (LVEF <45% on echocardiography or equivalent of MUGA) even if full recovery has occurred
  * Atrial fibrillation with a ventricular rate of >100 beats per minute on ECG at rest
* Uncontrolled infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active primary immunodeficiency
* Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome, or renal tubular acidosis.
* Current gastrointestinal conditions such as refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of small bowel, symptomatic inflammatory bowel disease, or ulcerative colitis, or partial or complete bowel obstruction.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (colitis, Crohn's), celiac disease, systemic lupus erythematosus, Wegener syndrome, myasthenia gravis, Graves' disease, rheumatoid arthritis, uveitis.

The following exceptions are:

* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto's syndrome) stable on hormone replacement
* Psoriasis that does not require systemic therapy
* Patients with celiac disease that is controlled by diet alone

  • Ophthalmological conditions as follows:
* Current or past history of retinal vein occlusion
* Known intraocular pressure (IOP)>21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma.
* Subjects with ophthalmological findings secondary to long standing optic pathway glioma (such as visual loss, optic nerve pallor, or strabismus) or long standing orbito-temporal PN (such as vision loss, strabismus) will not be considered a significant abnormality for purposes of this study.

Any Supplementation with vitamin E.

Hypersensitivity to investigational products, or drugs with similar chemical structures to investigational products.

Patients unwilling or unable to comply with the protocol.

While not an exclusion criterion, unless clinically indicated, patients should avoid taking other additional non-study medications that may interfere with the study medications. In particular, participants should avoid medications that are known to either induce or inhibit the hepatic activity of CYP1A2, CYP2C19, and CYP3A4.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2031-05-15 (Estimated); Study Completion 2032-05-15 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability Selumetinib with ZEN-3694 | From first dose through the end of the first treatment cycle for each participant at each dose level (up to 28 days).
  To determine the safety, tolerability, and recommended doses of selumetinib given in combination with ZEN-3694 in participants with refractory sarcomas including MPNST.
  The Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of selumetinib in combination with ZEN-3694 will be determined based on dose-limiting toxicities (DLTs) observed during the first cycle of therapy. DLTs are defined as grade ≥3 toxicities attributable to the study drugs, assessed according to CTCAE v5. Dose escalation will proceed in cohorts of 3-6 participants, with possible dose de-escalation if ≥33% of participants experience a DLT. At the RP2D, the cohort may be expanded to up to six additional participants to further evaluate pharmacokinetics and tolerability.
Part B: Safety and Tolerability of Durvalumab with Combination of Selumetinib and ZEN-3694 | From first dose through the end of the first treatment cycle for each participant at each dose level (up to 28 days).
  To determine the safety, tolerability, and recommended doses of durvalumab when given in combination with selumetinib and ZEN-3694 in participants with refractory sarcomas including MPNST.
  The Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of the combination of selumetinib, ZEN-3694, and durvalumab will be determined based on dose-limiting toxicities (DLTs) observed during the first cycle of therapy. DLTs are defined as grade ≥3 toxicities attributable to the study drugs, assessed according to CTCAE v5. Dose escalation will proceed in cohorts of 3-6 participants, with possible dose de-escalation if ≥33% of participants experience a DLT. At the RP2D, the cohort may be expanded to up to six additional participants to further evaluate pharmacokinetics and tolerability.
Part C: Determine the Clinical Benefit of Selumetinib, ZEN-3694 and Durvalumab | From first dose through completion of 4 treatment cycles for each participant (up to 112 days).
  Clinical benefit rate defined as radiographic complete response, partial response, or stable disease, greater than or equal to four cycles.
  The primary endpoint is the clinical benefit rate, defined as the proportion of evaluable participants achieving a complete response (CR), partial response (PR), or stable disease (SD) for at least 4 treatment cycles. A Simon's optimal two-stage phase 2 design will be used to evaluate efficacy in participants with unresectable or metastatic NF1-associated MPNST. In the first stage, 9 participants will be enrolled; the trial will stop early if 0 participants respond. If the study continues to the second stage, a total of 17 participants will be enrolled, and the treatment will be considered ineffective if ≤2 participants respond. The target clinical benefit rate is 30% (p1 = 0.30), and a rate ≤5% (p0 = 0.05) is considered uninteresting.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No